CLINICAL TRIAL: NCT06178666
Title: A Feasibility Study of a Controlled Human Infection Model (CHIM) With Intradermal Bacillus Calmette-Guérin (BCG) Injection in Malawi
Brief Title: A Controlled Human Infection Model (CHIM) With Intradermal BCG in Malawi
Acronym: MLWBCGCHIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Liverpool School of Tropical Medicine, United Kingdom (Unknown); Fred Hutchinson Cancer Center (Other); University of Liverpool (Other); Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-Marvels-003; 23-083 (Other: Liverpool School Tropical Medicine)
Record Dates: First submitted 2023-12-07; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: A feasibility study of a controlled human infection model (CHIM) with intradermal bacillus Calmette-Guérin (BCG) injection in Malawi
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose of BCG being tested in dose ranging study (Experimental): The lowest dose of BCG (standard Malawi BCG vaccine (BCG Bulgaria 150000-600000 cfu) given as intradermal injection) will be used to determine safety and feasibility. The investigators do not expect to be able to meet study endpoints in this arm which will recruit 10 subjects.
  Interventions: Biological: BCG
- Mid-range dose BCG being tested in dose ranging study (Experimental): The mid-range dose of BCG (4x standard Malawi dose (BCG Bulgaria 600000-2400000 cfu intradermal) and equal to the model tested in Oxford, UK) will be used to determine safety and feasibility. The investigators hope to to be able to meet study endpoints (measuring microbiological and immunological features of BCG skin lesion) in this arm which will recruit 10 subjects.
  Interventions: Biological: BCG
- High dose BCG being tested in dose ranging study (Experimental): The highest dose of BCG (10x standard Malawi dose (BCG Bulgaria 2400000-9600000 cfu intradermal) and equal to USA dose used in Seattle) will be used to determine safety and feasibility. The investigators expect to be able to meet study endpoints in this arm which will recruit 10 subjects. In the event that study endpoints are met in the mid-range dose, the investigators will introduce a rifampicin dosing schedule to this arm.
  Interventions: Biological: BCG

INTERVENTIONS:
Biological: BCG — Three dose levels of intradermal BCG
  Other Names: Bacille Calmette Guerin

SUMMARY:
Despite tremendous efforts, an effective tuberculosis (TB) vaccine remains elusive. TB continues to infect and kill many. In 2021, TB infected more than 10 million and killed 1.6 million people. To date, the M.bovis bacille Calmette Guerin (BCG) is the only licensed vaccine against tuberculosis (TB). Efforts to come up with new and effective vaccines have not been successful. Partially, the lack of suitable disease models and protection correlates hinders the research of new vaccines. Controlled human infection model studies (CHIM) involve administering disease-causing microbes to healthy individuals, with continued monitoring of disease response. These studies have been used to study malaria, typhoid, pneumococcal pneumonia and the recent SARS-CoV-2 vaccines. The BCG-Controlled Human Infection Model (BCG-CHIM) will allow accurate dosing with safe mycobacteria as well as minimal tissue sampling to understand immunity to mycobacteria. Considering that the M. bovis BCG is a safe living Mycobacteria, it can be used as a CHIM against which to test new vaccines.

DETAILED DESCRIPTION:
Tuberculosis (TB) is a leading cause of death from a single infectious agent worldwide and is an acknowledged major challenge in Malawi. Globally in 2021, there were an estimated 10.6 million people unwell with TB and an estimated 1.6 million deaths caused by TB. Furthermore, the global TB incidence could be accelerated to an average of 17% per year between 2025 and 2035 owing to the disruption to TB services caused by the COVID pandemic. TB diagnosis is challenging, and drug treatment can be prolonged, harmful, costly, and complex, especially in the increasingly common context of drug resistant M. tuberculosis. For these reasons an effective vaccine to prevent disease is a global public health priority, and drugs to allow shorter courses of effective therapy are urgently needed.

At present, the only licensed vaccine is the bacille Calmette-Guérin (BCG) vaccine (BCG Bulgaria is the Malawi licensed strain). BCG has been administered globally to several billion people over the last 100 years and it has been part of the expanded program on immunisations since the early-1970s. BCG is effective in preventing disseminated TB disease, including tuberculous meningitis in childhood. However, it does not protect against pulmonary TB in many parts of the world, especially in the tropics where the incidence of TB is at its greatest. Since pulmonary TB is associated with the highest morbidity and mortality, the need to develop an effective vaccine against this disease is paramount, especially in Malawi where BCG protection is known to be minimal.

There are several novel vaccines for TB in clinical development, the most clinically advanced of which is M72/AS01E. The evaluation of candidate TB vaccines is challenging, and progress in the field is hampered by the lack of an immunological correlate of protection. Most routinely administered vaccines generate a quantifiable antibody response that correlates strongly with protection. In contrast, protection against TB is critically dependent on the cellular immune response, in particular CD4+ and also probably CD8+ T cell mediated cellular responses. The mechanisms of these responses are not fully understood .

Currently, to assess vaccine efficacy against TB there is no alternative to large randomized controlled trials. These efficacy trials for novel TB vaccines are difficult, long and very costly. For this reason, there is an urgent need for a valid, reliable, and strong evaluation technique to help distinguish between candidate TB vaccines' likely efficacy at Phase 3. Candidate vaccines which have passed successfully through phase I trials and are in Phase 2b efficacy studies could be included in human challenge protocols which could be designed to either measure prevention of infection (POI) or immunological endpoints. This would allow vaccine discovery to accelerate in a cost-effective manner. Similarly, successful development of new, safe and effective TB therapies face multiple challenges. A responsive controlled human infection model of TB infection could accelerate the development of new drugs and promote refinement of drug combination regimens.

Controlled human infection models (CHIMs) provide insight into disease pathogenesis and correlates of immune protection to support the development of novel vaccines.

The Malawi Liverpool Wellcome Trust has extensive experience of delivering CHIM studies in Malawi with Streptococcus pneumoniae and established technology transfer processes with previous successful transfer of the experimental human pneumococcal carriage model from Liverpool to Blantyre, Malawi. Before the Malawi BCG study, the team will also confirm feasibility of this established BCG model in Liverpool. The Liverpool team will be able to share techniques and expertise and compare data as the Liverpool population will have a different experience of BCG and tuberculosis in the community and are likely to show different results. A TB CHIM established in both the UK and Malawi has the potential to rapidly advance development of vaccines and therapeutics fit for use in populations that need them most.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-50 (inclusive)
* Resident near QECH, Blantyre (<1 hour drive) for the duration of the study period
* Allows the investigators to review the volunteer's medical history in the health passport book.
* Females of childbearing potential with a negative urine pregnancy test at screening and willing to practice adequate birth control measures during the study.
* Fluent spoken English or Chichewa - to ensure a comprehensive understanding of the research project and their proposed involvement.
* Capacity to provide informed consent before joining the study.
* Able and willing (in the investigators opinion) to comply with all the study requirements.

Exclusion Criteria:

* Laboratory evidence at screening of subclinical M. tb infection as indicated by a positive ELISPOT response to ESAT-6 or CFP-10 antigens. Volunteers discovered to have evidence of latent M. tb infection as defined by a positive ELISPOT test will be referred to the chest clinic for investigation for tuberculosis according to Malawi standard protocols.
* Clinical, radiological, or laboratory evidence of current active TB disease
* Clinically significant history of skin disorder, allergy, immunodeficiency (including HIV), cancer, cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness, or psychiatric disorder.
* Current medical issues. Volunteers who are excluded from the study because they have been discovered to have a previously undiagnosed condition thought to require further medical attention will be referred appropriately to QECH specialist services for further investigation and treatment.
* Acute respiratory tract infection in the four weeks preceding recruitment
* Any uncontrolled medical or surgical condition at the discretion of the study doctor
* Female participants who are pregnant, or intending to become pregnant, lactating or who Female participants who are unable to take contraception measures during the study.
* Smoking: Current (defined as ≥5/week) or ex-smoker (cigarettes / cigars / smoking of recreational drugs) in the last 6 months. Previous significant smoking history (more than 20 cigarettes per day for 20 years or the equivalent [>20 pack years]).Current alcohol and recreational drug use
* Regularly drinks ≥3units/day (male) or ≥2units/day (female)
* Uses recreational drugs.
* Participants may be excluded at the discretion of the research clinician.
* Concurrent oral or systemic steroid medication or the concurrent use of other immunosuppressive agents
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the challenge agent.
* Has received any vaccination within one month of screening visit.
* Any abnormality of screening blood or urine tests that is deemed to be clinically significant or that may compromise the safety of the volunteer in the study.
* Current involvement in another trial that involves regular blood tests or an investigational medicinal product.
* Use of an investigational medicinal product or non-registered drug, live vaccine, or investigational medical device for four weeks prior to dosing with the study challenge agent
* Participants who meet STOP criteria at the time of screening (see table 4)
* Any other issue which, in the opinion of the study staff, may
* Put the participant or their contacts at risk because of participation in the study,
* Adversely affect the interpretation of the study results, or
* Impair the participant's ability to participate in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Culture and PCR ascertainment of BCG load | 14 days
  BCG will be quantified in 4mm skin punch biopsy

SECONDARY OUTCOMES:
Immunological response to BCG | 14 days
  Innate, humoral and cellular immune functions will be quantified in 4mm skin punch biopsy, mucosal and blood samples using ELISA, flow cytometry, 10X single cell and geospatial transcriptomics.

OTHER OUTCOMES:
Microbiology and immunology | Day 2, 7, 14, 21, 28
  The BCG infection quantified in Outcome 1 will be compared with the Immunology determined in Outcome 2 to provide associations which may later be tested as correlates of protection.
Lung cellular and humoral immune response | Day 14 after inoculation
  Bronchoalveolar lavage will be collected in a subset of volunteers willing to undergo this procedure. Bronchoalveolar lavage cells will be studied by flow cytometry for phenotype and antigen specific cytokine production. BAL fluid will be used to measure anti-BCG Ig responses by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gordon, MD, Principal Investigator — Malawi Liverpool Wellcome Programme
Locations (1):
- Queen Elizabeth Central Hospital, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: No
Anonymised data will be shared in an online database. IPD would breach data protection guidelines and will not be necessary to interpret the study.

REFERENCES:
- [Background] Lin LL, Prow TW, Raphael AP, Harrold Iii RL, Primiero CA, Ansaldo AB, Soyer HP. Microbiopsy engineered for minimally invasive and suture-free sub-millimetre skin sampling. F1000Res. 2013 May 2;2:120. doi: 10.12688/f1000research.2-120.v2. eCollection 2013. PMID 24627782
- [Background] Lei BUW, Yamada M, Hoang VLT, Belt PJ, Moore MH, Lin LL, Flewell-Smith R, Dang N, Tomihara S, Prow TW. Absorbent Microbiopsy Sampling and RNA Extraction for Minimally Invasive, Simultaneous Blood and Skin Analysis. J Vis Exp. 2019 Feb 21;(144). doi: 10.3791/58614. PMID 30855573